CLINICAL TRIAL: NCT02117440
Title: Using Functional Image and Circulating Molecular Markers to Predict Tumor Control and Thoracic Toxicity in Treatment of Lung Cancer
Brief Title: Functional Image and Molecular Markers to Predict Treatment Outcomes in Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Lautenschlaeger, Assistant Professor of Radiation Oncology, Indiana University
Other Study IDs: IUSCC-0596; GRU CC-13-24C (Other: Georgia Regents University)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Lung Neoplasms
Keywords: Lung Cancer; Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buffy coat, plasma and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to apply various scans such as functional imaging, Fluorodeoxyglucose_Positron Emission Tomography (FDG-PET), 62Cu-ETS (Copper) PET, Ventilation/Perfusion Single Photon Emission Computerized Tomography (V/Q SPECT), cardiac magnetic resonance imaging (MRI), Tc-99m HMPAO SPECT/CT, and pulmonary function tests before, during and after treatment to see if it predicts how well the treatment works for your cancer and how well your lungs function during treatment. A Computerized Tomography (CT) will also be performed along with both of these procedures to help the researchers see clearly where your cancer or your healthy lung is located. The researchers also perform blood tests in this study to look for markers in your blood to see if it helps them determine your risk of developing side effects from radiation to the lungs. They will also measure your health-related quality of life before, during and after treatment. The researchers hope that this study will help them in the future to design radiation treatment plans that provide the best treatment for each individual patient.

DETAILED DESCRIPTION:
Primary aims:

1. To determine if tumor metabolic activity plus volume measured by 18F-FDG PET/CT and tissue/tumor perfusion measured by 62Cu-ETS-PET before and during treatment predicts CT tumor response 3 months after completion of treatment and 1 and 2 year local-regional progression-free survival.
2. To determine if functional imaging based lung dose-volume histograms (DVH) more accurately predict changes in diffusion capacity of lung for carbon monoxide (DLCO) compared to the DVH based on simulating CT. Degree of lung toxicity will also be documented by functional scans such as Tc-99m HMPAO imaging.
3. To determine if baseline level, or changes in blood markers such as TGFß1 measured during the course of radiation, predict changes in DLCO.

ELIGIBILITY:
Potentially eligible patients include all patients with stage I to IV lung cancer. Patient cannot have started systemic treatments or radiation treatments prior to enrollment on the study. Informed consent will be obtained in writing prior to initiating the study using a consent form approved by the local IRB.

Inclusion criteria

* Histologically confirmed lung cancer, or clinically diagnosed lung cancer.
* AJCC stage I to IV lung cancer requiring radiation therapy (3D conformal or stereotactic) or systemic therapy, with or without surgery.
* Patients participating treatment trials including targeted therapy, experimental therapy or immunotherapy are also eligible.
* Patients with a locoregional tumor recurrence following surgery will be eligible provided they meet other eligibility criteria.
* Patients must be 18 years of age or older and able to lie flat to obtain the functional scans or have blood access for blood samples
* Female patients with reproductive capability must be willing to use effective contraception.
* Patients must be willing and able to be compliant with all procedures and visits required for this protocol (pre-treatment, during treatment, and optionally throughout follow-up period).
* Patients must sign an informed consent form for study.
* Patients must be willing and able to adhere to a special low-carb diet 24-48 hours prior to and fast 8-12 hours prior to every 18F-FDG PET scan

Exclusion criteria

* Pregnancy if the patient is receiving radiation therapy
* Lactation if the patient is receiving radiation therapy
* Patients with diabetes mellitus, with uncontrolled fasting blood glucose level (above 200 mg/dl)
* Inability to lie flat for the duration of PET/CT and V/Q SPECT/CT (approximately 45 minutes for each study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Investigate predictive models for long-term tumor control and late treatment lung toxicity by using FDG-PET-CT, V/Q SPECT-CT and blood test during the course of radiation therapy. | Up to 5 years after radiation completion
  Investigate predictive models for long-term tumor control and late treatment lung toxicity by using FDG-PET-CT, V/Q SPECT-CT and blood test during the course of radiation therapy. As secondary analysis, demographic and baseline clinical variables will be added to the model to determine if they add predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Kong, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States